CLINICAL TRIAL: NCT04877379
Title: VNRX-7145-102: A Randomized, Drug-Drug Interaction Study to Assess the Safety and Pharmacokinetics (PK) of VNRX-7145 and VNRX-5024 (Ceftibuten) in Healthy Adult Volunteers
Brief Title: VNRX-7145 Drug-Drug Interaction in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-7145-102; 272201600029C-P00007-9999-2 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ceftibuten

STUDY DESIGN:
Intervention Model Description: Part 1: Crossover Parts 2&3: Parallel
Who Masked: Participant, Investigator
Masking Description: Part 1: Unblinded Parts 2&3: Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 (Experimental): Subjects will receive single doses of VNRX-7145 or VNRX-5024 alone and in combination. All subjects will receive study drug in the sequence specified by the randomization schedule.
  Interventions: Drug: VNRX-7145; Drug: VNRX-5024 (ceftibuten)
- Part 2A (Experimental): Multiple dose administration of VNRX-7145 q8h for 10 days
  Interventions: Drug: VNRX-7145
- Part 2B (Placebo Comparator): Multiple dose administration of placebo q8h for 10 days
  Interventions: Drug: Placebo
- Part 3A (Experimental): Multiple dose administration of low dose VNRX-7145 + VNRX-5024
  Interventions: Drug: VNRX-7145; Drug: VNRX-5024 (ceftibuten)
- Part 3B (Experimental): Multiple dose administration of high dose VNRX-7145 + VNRX-5024
  Interventions: Drug: VNRX-7145; Drug: VNRX-5024 (ceftibuten)
- Part 3C (Placebo Comparator): Multiple dose administration of Placebo (matching VNRX-7145 + VNRX-5024)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VNRX-7145 — β-lactamase inhibitor
  Arms: Part 1; Part 2A; Part 3A; Part 3B
Drug: VNRX-5024 (ceftibuten) — β-lactam antibiotic
  Arms: Part 1; Part 3A; Part 3B
Drug: Placebo — Placebo
  Arms: Part 2B; Part 3C

SUMMARY:
This study will provide an initial assessment of the safety and PK of VNRX-7145 and VNRX-5024 (ceftibuten) when administered as single agents and with co-administration in a single dose cross-over design in Part 1. In Part 2, subjects will receive 500 mg of VNRX-7145 or matching placebo q8h for 10 days. VNRX-7145 and VNRX-5024 (ceftibuten) will be administered every 8 hours (q8h) for 10 days at 2 dose levels of VNRX-7145 in Part 3.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-55 years
2. Males or non-pregnant, non-lactating females
3. Body mass index (BMI): ≥18.5 kg/m2 and ≤32.0 kg/m2
4. Normal blood pressure
5. Normal lab tests

Exclusion Criteria:

1. History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorders
2. History of drug allergy or hypersensitivity to penicillin, cephalosporin, or beta-lactam antibacterial drug
3. Use of antacid medications
4. Abnormal ECG or history of clinically significant abnormal rhythm disorder
5. Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Cmax | 0-48 hours
  concentration time data
Part 1: AUC0-inf | 0-48 hours
  Area under the concentration-time curve from time-zero extrapolated to infinity based on collected PK
Parts 2&3: Number of subjects with adverse events | Day 15 (+2)

SECONDARY OUTCOMES:
Part 1: Number of subjects with adverse events | Day 14 (+2)
Parts 2&3: AUC0-tau | Day 1
Parts 2&3: AUC0-tau | Day 10
Parts 2&3: Cmax | Day 1
Parts 2&3: Cmax | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- PRA Health Sciences - Early Development Services, Groningen, Netherlands

REFERENCES:
- [Derived] de Oliveira CF, Dorr MB, van de Wetering J, Lowe K, Sabato P, Winchell G, Chen H, McGovern PC. Safety and pharmacokinetics of single and multiple doses of ledaborbactam etzadroxil with or without ceftibuten in healthy volunteers. Antimicrob Agents Chemother. 2025 Sep 3;69(9):e0021025. doi: 10.1128/aac.00210-25. Epub 2025 Aug 5. PMID 40762486